CLINICAL TRIAL: NCT05728242
Title: Perioperative Point-of-care Gastric Ultrasound for Surgical Fracture Repair: Effect of Stress on Gastric Emptying
Brief Title: Point-of-care Gastric Ultrasound for Fracture Surgery
Status: Recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 142-2021
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-06

CONDITIONS: Pneumonia, Aspiration; Gastric Content; Fractures, Bone
Keywords: gastric ultrasound; aspiration pneumonia; gastric emptying; fracture surgery
MeSH Terms: conditions — Pneumonia, Aspiration; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gastric ultrasound — Preoperative gastric antrum examination to detect gastric content (empty, liquid, or solid) and measure gastric volume

SUMMARY:
Although there are fasting guidelines offered by the American Society of Anesthesiology (ASA) for managing preoperative patient assessment, some patients may need to be more cautious about the risk of aspiration. Since ultrasound has been a part of perioperative anesthesiology practice, it is simple to assess gastric content preoperatively with bedside ultrasonography (USG). More research is necessary to define elective surgeries with a possible risk of aspiration. Therefore, we aimed to evaluate the adequacy of standard fasting protocols in post-traumatic fracture surgery by measuring and evaluating gastric volume and content with USG in the preoperative operating room.

DETAILED DESCRIPTION:
Pulmonary aspiration of the gastric content is an avoidable complication that can lead to severe morbidity and even mortality. Although there are fasting guidelines offered by the American Society of Anesthesiology (ASA) for managing preoperative patient assessment, some patients may need to be more cautious about the risk of aspiration. Patients with gastrointestinal disorders or diabetes and conditions like pregnancy and obesity have been assessed because of possible delayed gastric emptying. Besides children, elderly and acute traumatic events have also been evaluated since they may not obey or fulfill preoperative fasting rules. Since ultrasound has been a part of perioperative anesthesiology practice, it is simple to assess gastric content preoperatively with bedside ultrasonography (USG). It may be logical to standardize gastric USG principally in situations concluding in decreased gastric peristalsis and gastric emptying. More research is necessary to define elective surgeries with possible risks.

Although recent studies have investigated the effect of gastric USG on risk stratification and clinical decision-making, especially in patients with special conditions, an investigation on patients scheduled for fracture surgery has not been evaluated. It is known that there is an inflammation process that extends up to the 4th day of trauma and an increase in stress hormones in fractures. Therefore, we aimed to evaluate the adequacy of standard fasting protocols in post-traumatic fracture surgery by evaluating gastric volume and content with USG in the preoperative operating room.

Material and Method Study design and study subjects The study was designed as prospective observational research after approval of our Institutional ethics committee (dossier no:142-2021) and planned to allocate at least 50 patients after obtaining written informed consent. Patients over 18 with the American Society of Anesthesiology (ASA) I-III who are scheduled for orthopedic surgery within three days after fracture are eligible for this study. Exclusion criteria are conditions or diseases affecting gastric emptying and peristalsis: body mass index over 35; gastroesophageal reflux disease; diabetes mellitus; esophageal abnormalities; history of gastric surgery; gastric or peptic ulcus; pregnancy; preoperative narcotic analgesic usage; connective tissue disorders like scleroderma or amyloidosis; hiatal hernia; gallbladder and choledochal stone.

Anesthesia, intervention, and post-interventional follow-up Patients are questioned about their fasting status; content and timing of the last food or drink. The attending anesthesiologist notes the decided anesthesia plan before intervention. An ultrasound examination is performed by another anesthesiologist, experienced with ultrasound at least for 5 years and all evaluations will be done by the same anesthesiologist. Gastric volume is investigated first in the supine and the right lateral decubitus position (RLD). Both qualitative (nature of gastric content) and quantitative (volume of gastric fluid) measurements are used to conclude the amount of gastric content and aspiration risk. For assessment 3 grade system will be used as described by Perlas. Grade 0, no gastric content within the antrum at both positions; Grade 1, gastric content is seen only at the RLD position; Grade 2 gastric content was detected in both positions. If gastric content is detected then, quantitive assessment is established by measuring antral area (Antral cross-sectional area = anterior-posterior diameter (D1) × craniocaudal diameter (D2) × π/4) and total gastric volume will be calculated with the formula (gastric volume (mL) = 27.0 + 14.6 x right-lat CSA - 1.28 x age). If the total gastric volume is over 1,5 ml /kg, grade 2; if 1,5- 0,8 ml/kg, grade 1; ˂ 0,8 ml/kg will be noted as grade 0. Finally, if the patient is considered to be grade 2, it will be evaluated as high aspiration risk, and if the anesthesia plan needs to be changed, it will be recorded as well. For patients concluded to have grades 1 and 2, postoperative follow-up will search for nausea and vomiting, fever, cough, tachypnea, and tachycardia within 48 hours. If any of these have occurred, aspiration pneumonia will be searched with further examination or imagination.

ELIGIBILITY:
Inclusion Criteria:

* • American Society of Anesthesiologists (ASA) Physical Status classification I to III

  * Patients necessitating surgery after traumatic fracture

Exclusion Criteria:

* • Patients with a body mass index over 35

  * Diseases that may lead to gastroparesis (
  * Known gastroesophageal reflux disease
  * Known autonomic neuropathy
  * Known diabetes mellitus
  * Known or operated esophageal abnormalities
  * History of gastric surgery
  * Acute gastric or peptic ulcus
  * Pregnancy
  * Preoperative narcotic analgesic usage
  * Known connective tissue disorders like scleroderma or amyloidosis
  * Known hiatal hernia
  * Known gallbladder and choledochal stone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been admitted to fracture surgery within 3 days of the trauma
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
gastric volume(ml) | preoperative, only one measurement
  gastric volume calculated with gastric volume (mL) = 27.0 + 14.6 x right-lat CSA - 1.28 x age and Antral cross-sectional area = anterior posterior diameter (D1) × cranio-caudal diameter (D2) × π/4 . Evaluation is done as over 1,5 ml /kg grade 2; if 1,5- 0,8 ml/kg, grade 1; ˂ 0,8 ml/kg, grade 0
gastric content | preoperative, only one examination
  Grade 0, no gastric content within the antrum at both positions ( supine and right lateral decubitis(RLD)); Grade 1, gastric content is seen only at RLD position; Grade 2 gastric content was detected in both positions

SECONDARY OUTCOMES:
nausea or vomiting | postoperative 24 hour
  postoperative nausea or vomiting
aspiration pneumonia | postoperative 48 hours
  fever, cough, tachypnea, tachycardia within and if there is any of these has occured, aspiration pneumonia will be searched with further examination or imagination for certain diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Principal Investigator — Haseki Training and Research Hospital Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alakkad H, Kruisselbrink R, Chin KJ, Niazi AU, Abbas S, Chan VW, Perlas A. Point-of-care ultrasound defines gastric content and changes the anesthetic management of elective surgical patients who have not followed fasting instructions: a prospective case series. Can J Anaesth. 2015 Nov;62(11):1188-95. doi: 10.1007/s12630-015-0449-1. Epub 2015 Aug 4. PMID 26239668
- [Result] Zhang G, Huang X, Shui Y, Luo C, Zhang L. Ultrasound to guide the individual medical decision by evaluating the gastric contents and risk of aspiration: A literature review. Asian J Surg. 2020 Dec;43(12):1142-1148. doi: 10.1016/j.asjsur.2020.02.008. Epub 2020 Mar 11. PMID 32171605